CLINICAL TRIAL: NCT01063023
Title: Effect of BMS-650032 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate (Ortho Tri- Cyclen (R)) in Healthy Female Subjects
Brief Title: Drug Interaction Oral Contraceptive Pill (OCP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AI447-019
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — norgestimate, ethinyl estradiol drug combination; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A - Ortho Tri-Cyclen® (Active Comparator): 1 to 28 days
  Interventions: Drug: Ortho Tri-Cyclen®
- Arm B - Ortho Tri-Cyclen® (Active Comparator): 29 to 56 days
  Interventions: Drug: Ortho Tri-Cyclen®
- Arm C - Ortho Tri-Cyclen® + BMS-650032 (Active Comparator): Ortho Tri-Cyclen®: 57 to 77 days
  BMS-650032: 68 to 77 days
  Interventions: Drug: Ortho Tri-Cyclen®; Drug: BMS-650032

INTERVENTIONS:
Drug: Ortho Tri-Cyclen® — Tablets, Oral, 1 Tablet, once daily
Drug: BMS-650032 — Tablets, Oral, 600 mg, BID
  Arms: Arm C - Ortho Tri-Cyclen® + BMS-650032

SUMMARY:
To assess the effects of BMS-650032 on Pharmacokinetics (PK) of ethinyl estradiol (EE) and norelgestromin (NGMN) in healthy female subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females, 18-40 years, BMI 18 - 32kg/m². Must use an acceptable method of contraception to avoid pregnancy throughout the study and 8 weeks after last dose of study drug

Exclusion Criteria:

* Abnormal pap smear within 1 year prior to day 1
* Any significant or chronic uncontrolled medical illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters for ethinyl estradiol (EE), norelgestromin (NGMN) and norgestrel (NG), AUC (TAU) | 24 hours of dosing

SECONDARY OUTCOMES:
To assess the safety and tolerability of investigational drug and Ortho Tri-Cyclen® when administered | Safety will be assessed through day 78
To characterize the PK of norgestrel when Ortho Tri-Cylen® is administered alone and in combination | PK assessments will be done on Day 49, 50, 77 and 78

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pra International, Lenexa, Kansas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx